CLINICAL TRIAL: NCT04451252
Title: Observational Prospective Single Centre Study of the Response to Interventional Pain Management Techniques in Chronic Low Back Pain in Adults. 1 and 6 Months Follow-up. Multivariate Analysis of Predictors of Response. Predictive Model.
Brief Title: Predicting Response to Interventional Pain Management Techniques in Chronic Low Back Pain in a Prospective Cohort.
Acronym: PReTI-Back
Status: Completed | Type: Observational
Sponsor: Santiago Garcia-Hernandez (Other)
Responsible Party: Sponsor-Investigator, Santiago Garcia-Hernandez, Aneaesthesiology, Critical Care and Pain Medicine Resident Trainee. Hospital General Universitario Gregorio Marañon., Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: PRETI-DOL-V1
Record Dates: First submitted 2020-06-15; First posted 2020-06-30 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Low Back Pain; Pain Measurement; Chronic Pain; Analgesia, Epidural; Clinic, Pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Agnosia; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Fluoroscopically guided lumbar medial branch nerve radiofrequency denervation. — While in prone position, lumbar facet joints are identified by fluoroscopy. 18 gauge needles are then advanced aiming to the medial branch of lumbar facet joints. Correct positioning is confirmed by anteroposterior and lateral fluoroscopy. Then, the needles are attached to the radiofrequency device. Correct positioning of the needles is confirmed also by sensitive stimulation (paresthesia evocation) with the following settings: 50 Hz (hertz), 1ms, 0,6V (volts). In order to avoid motor lesion, it is confirmed that no motor response is produced with 2Hz, 2ms (millisecond) and twice the voltage that produced sensitive response. After correct positioning and repositioning the needles if needed, conventional radiofrequency ablation of medial branch nerves is performed using the following settings: 90 seconds, 80º Celsius degrees.
  The selection of target facet joints is made based on clinical findings. Some patients receive bilateral while other unilateral facet joint denervation.
Procedure: Fluoroscopically guided lumbar medial branch nerve injection. — While in prone position, lumbar facet joints are identified by fluoroscopy. An anteroposterior image of the lumbar vertebrae is obtained. Then, the fluoroscope is tilted between 10 to 20 degrees to the side to inject. 22 gauge needles are then advanced aiming to the medial branch of lumbar facet joints.
  The selection of target facet joints is made based on clinical findings. Some patients receive bilateral while other unilateral facet joint denervation. Correct positioning is confirmed with anteroposterior and lateral fluoroscopy. A mixture of 3 ml of ropivacaine 0,2% + 1 ml (40 mg) of triamcinolone (trigon depot) is prepared. 1 ml of the mixture is injected in each lumbar facet joint through the needles. Four facet joints are selected for therapy. Some patients receive bilateral and other unilateral but contiguous medial branch nerve injection.
Procedure: Fluoroscopically guided lumbar epidural corticosteroid injection. — With the patient in prone position and guided by fluoroscopy, an epidural needle attached to a syringe filled with saline serum is advanced through the interlaminar approach using a loss of resistance technique for the identification of the lumbar epidural space. When loss of resistance is encountered, 1 ml of iodinated contrast is injected. After fluoroscopical confirmation of epidural spilling, a mixture of 4 ml of ropivacaine 0,1%, 2 ml (12 mg) of betamethasone and 2 ml of saline serum is injected in the epidural space. The lumbar level to which it infiltrates depends on each patient.
Procedure: Fluoroscopically guided caudal epidural corticosteroid injection. — With the patient in prone position and guided by fluoroscopy, an epidural needle attached to a syringe filled with saline serum is advanced through the sacral hiatus using a loss of resistance technique for the identification of the epidural space. When loss of resistance is encountered, 2 ml of iodinated contrast is injected. After fluoroscopical confirmation of epidural spilling, a mixture of 7 ml of ropivacaine 0,2%, 2 ml (12 mg) of betamethasone and 7 ml of saline serum is injected in the epidural space.
Procedure: Fluoroscopically guided pulsed radiofrequency of the lumbar dorsal root ganglion. — With the patient in prone position and guided by fluoroscopy, a 18 gauge needle is advanced aiming to the intervertebral foramen. Patient is cautioned about the paresthesia which will be felt. A lateral view was taken occasionally to confirm position. 0.5 ml of iodinated contrast is injected to confirm the position of the needle. Then 1 ml of the combination of 12mg of betamethasone and 1ml of ropivacaine 0.2% is injected over the affected root. Then, the needle is attached to the radiofrequency device. Correct positioning of the needles is confirmed also by sensitive stimulation (paresthesia evocation) with the following settings: 50 Hz, 1ms, 0,6V. In order to avoid motor lesion, it is confirmed that no motor response is produced with 2Hz, 2ms and twice the voltage that produced sensitive response. After correct positioning is confirmed, pulsed radiofrequency ablation of lumbar dorsal root ganglion is performed using the following settings: 4 minutes, 42ºC (degrees Celsius).
Procedure: Fluoroscopically guided transforaminal epidural corticosteroid injection or lumbar selective root block. — With the patient in prone position and guided by fluoroscopy, a 22 french needle is then advanced aiming to the intervertebral foramen. Patient is cautioned about the paresthesia which will be felt along the course of the lumbar root when the needle touches the nerve. A lateral view was taken occasionally to confirm position. 0.5 ml of iodinated contrast is injected to confirm the position of the needle. Then 1 ml of the combination of 12mg of betamethasone and 1ml of ropivacaine 0.2% is injected over the affected root.

SUMMARY:
The main aim of this study is to identify factors that may be associated with a better or worse response to interventional pain management therapies for the treatment of chronic lumbar pain in adult patients. If several predictive factors are to be identified, a predictive model will be developed.

DETAILED DESCRIPTION:
Chronic lumbar pain is a common affection in the adult population, and an important source of chronic incapacity and impaired quality of life. There is a wide range of therapeutic options for the treatment of chronic lumbar pain. This study will analyze the response to several interventional pain management techniques and will search for factors that may be associated to a better or worse response to the techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old with chronic lumbar pain to whom one of the following interventional pain management techniques has been indicated:
* Radiofrequency lumbar facet joint injection
* Radiofrequency lumbar facet joint denervation
* Lumbar epidural corticosteroid injection
* Caudal epidural corticosteroid injection
* Pulsed radiofrequency of the lumbar dorsal root ganglion
* Dorsal root ganglion injection

Exclusion Criteria:

* Patients that have not undergone the interventional pain management technique. The interventional pain management technique is considered not performed if it is not done after a twelve month period after recruitment.
* Patients who are not willing to participate.
* Patients of whom it is impossible to obtain data of response.
* Patients who undergo low back surgery while they are in the study.
* Patients who suffer from an intercurrent disease that may interfere with the evaluation of chronic lumbar pain.
* Patients who suffer from myofascial pain syndromes.
* Patients who undergo pulsed radiofrequency denervation for the treatment of sacroiliac joint syndrome.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population consist of adult outpatients with chronic low back pain in the Chronic Pain Unit of our University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-07-04 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical response to IPMT after 4 weeks follow-up after the IPMT is performed (composite outcome) | Baseline (prior to the Interventional Pain Management Therapy); Week 4 after IPMT
  Clinical response after 4 week follow-up is going to be defined as composite outcomes:
  * Positive strong response (PSR-4W): a positive strong response to the interventional pain management therapy after 4 weeks follow-up is defined as a composite outcome. Patients must meet both the following criteria:
    * A decrease in Numeric Rating Scale of at least 3 points.
    * A decrease in the Oswestry Disability Index of al least 40%.
  * Positive moderate response (PMR-4W): a positive moderate response to the interventional pain management therapy after 4 weeks follow-up is defined as a composite outcome. Patients must meet both the following criteria:
    * A decrease in Numeric Rating Scale of at least 2 points.
    * A decrease in the Oswestry Disability Index of al least 20%.
  * No response (NR-4W): no response to IPMT after 4 weeks follow-up is defined as those patients not included in either of the previous categories.
Factors that may be associated with no response to the IPMT at 4 weeks follow-up. | Response will be measured after 4 weeks follow-up after the IPMT.
  14 candidate variables will be analyzed for association to no response to the IPMT at 4 weeks (NR-4W). All the variables are qualitative, dichotomic, yes/no:
  1. Work sick leave.
  2. Depression/Anxiety.
  3. Obesity.
  4. Existence of another chronic pain.
  5. Failed back surgery syndrome.
  6. Radicular compression in imaging.
  7. Herniated disc in imaging.
  8. Radiate pain.
  9. Age: older than 65 years old (>65 years old).
  10. Chronic therapy with opioid medication.
  11. Chronic therapy with gabapentionids.
  12. Chronic therapy with opioid medication AND gabapentinoids.
  13. Clinical Frailty Scale >3 (≥4).
  14. Initial Oswestry Disability Index ≥40.
Factors that may be associated with a positive response to the IPMT (PSR-4W or PMR-4W). | Response will be measured after 4 weeks follow-up.
  14 candidate variables will be analyzed for association to PSR-4W or PMR-4W to the IPMT at 4 weeks. All the variables are qualitative, dichotomic, yes/no:
  1. Working.
  2. Depression/Anxiety.
  3. Obesity.
  4. Failed back surgery syndrome.
  5. Radicular compression in imaging.
  6. Herniated disc in imaging.
  7. Radiate pain.
  8. Age: younger than 45 years old (<45 years old).
  9. Chronic therapy with opioid medication.
  10. Chronic therapy with gabapentinoids medication.
  11. Chronic therapy with opioid medication AND gabapentinoids.
  12. Clinical Frailty Scale <3.
  13. Initial Oswestry Disability Index ≥40.
  14. Subjective good subjective result in previous performed interventional pain management therapies.
Clinical response to IPMT after 24 weeks follow-up after the IPMT is performed (composite outcome). | Response will be measured after 24 weeks follow-up after the IPMT.
  Clinical response after 24 week follow-up is going to be defined as composite outcomes:
  * Positive strong response (PSR-24W): a positive strong response to the interventional pain management therapy after 24 weeks follow-up is defined as a composite outcome. Patients must meet both the following criteria:
    * A decrease in Numeric Rating Scale of at least 3 points.
    * A decrease in the Oswestry Disability Index of al least 40%.
  * Positive moderate response (PMR-24W): a positive moderate response to the interventional pain management therapy after 24 weeks follow-up is defined as a composite outcome. Patients must meet both the following criteria:
    * A decrease in Numeric Rating Scale of at least 2 points.
    * A decrease in the Oswestry Disability Index of al least 20%.
  * No response (NR-24W): no response to IPMT after 24 weeks follow-up is defined as those patients not included in either of the previous categories.
Factors that may be associated with no response to the IPMT at 24 weeks follow-up. | The factors will be recorded at baseline; the response will be measured at after 24 weeks follow-up.
  14 candidate variables will be analyzed for association to no response to the IPMT at 24 weeks (NR-24W). All the variables are qualitative, dichotomic, yes/no:
  1. Work sick leave.
  2. Depression/Anxiety.
  3. Obesity.
  4. Existence of another chronic pain.
  5. Failed back surgery syndrome.
  6. Radicular compression in imaging.
  7. Herniated disc in imaging.
  8. Radiate pain.
  9. Age: older than 65 years old (>65 years old).
  10. Chronic therapy with opioid medication.
  11. Chronic therapy with gabapentinoids medication.
  12. Chronic therapy with opioid medication AND gabapentinoids.
  13. Clinical Frailty Scale >3 (≥4).
  14. Initial Oswestry Disability Index ≥40.
Factors that may be associated with a positive response to the IPMT after a 24 weeks follow-up (PSR-24W or PMR-24W). | Response will be measured after 24 weeks follow-up after the IPMT.
  14 candidate variables will be analyzed for association to PSR-4W or PMR-4W to the IPMT at 24 weeks. All the variables are qualitative, dichotomic, yes/no:
  1. Working.
  2. Depression/Anxiety.
  3. Obesity.
  4. Failed back surgery syndrome.
  5. Radicular compression in imaging.
  6. Herniated disc in imaging.
  7. Radiate pain.
  8. Age: younger than 45 years old (<45 years old).
  9. Chronic therapy with opioid medication.
  10. Chronic therapy with gabapentinoids medication.
  11. Chronic therapy with opioid medication AND gabapentinoids.
  12. Clinical Frailty Scale <3.
  13. Initial Oswestry Disability Index ≥40.
  14. Good subjective result in previous performed interventional pain management therapies.

SECONDARY OUTCOMES:
Validation a predictive model for positive response to the IPMT after 4 weeks | Response will be measured after 4 weeks follow-up after the IPMT.
  In case that several predictive variables are identified, a predictive model will be developed, either for predicting good and/or bad response.
Validation a predictive model for positive response to the IPMT after 24 weeks | Response will be measured after 24 weeks follow-up after the IPMT.
  In case that several predictive variables are identified, a predictive model will be developed, either for predicting good and/or bad response.
Identifying other variables that may be associated with a good or bad response to an interventional pain management therapy (IPMT) at 4 weeks | Response will be measured after 4 weeks follow-up after the IPMT
  Other variables recorded in the Data Collection Logbook of our study will be analyzed looking for other associations:
  * Fibromyalgia.
  * Depression, anxiety and/or mixed axiety-depressive disorder.
  * Obesity.
  * Other chronic pain.
  * Failed back surgery syndrome.
  * Osteoporotic fracture.
  * Lumbar canal stenosis syndrome.
  * Irradiated pain to leg.
  * Diabetes Mellitus.
  * Arthrosis.
  * Inflammatory arthritis.
  * Oncologic condition.
  * Osteoporosis.
  * Substance abuse disorder.
Identifying other variables that may be associated with a good or bad response to an interventional pain management therapy (IPMT) at 24 weeks | Response will be measured after 24 weeks follow-up after the IPMT
  Other variables recorded in the Data Collection Logbook of our study will be analyzed looking for other associations:
  * Fibromyalgia.
  * Depression, anxiety and/or mixed axiety-depressive disorder.
  * Obesity.
  * Other chronic pain.
  * Failed back surgery syndrome.
  * Osteoporotic fracture.
  * Lumbar canal stenosis syndrome.
  * Irradiated pain to leg.
  * Diabetes Mellitus.
  * Arthrosis.
  * Inflammatory arthritis.
  * Oncologic condition.
  * Osteoporosis.
  * Substance abuse disorder.
Analyzing the response after 4 weeks to therapy of each interventional pain management therapy alone, and which variables may be associated with a better response to therapy. | Response will be measured after 4 weeks follow-up after the IPMT
  The therapies that will be analyzed are:
  * Fluoroscopically guided lumbar medial branch nerve radiofrequency denervation.
  * Fluoroscopically guided lumbar facet joint injection.
  * Fluoroscopically guided lumbar epidural corticosteroid injection.
  * Fluoroscopically guided caudal epidural corticosteroid injection.
  * Fluoroscopically guided pulsed radiofrequency of the lumbar dorsal root ganglion.
  * Fluoroscopically guided transforaminal epidural corticosteroid injection or lumbar selective root block.
Analyzing the response after 24 weeks to therapy of each interventional pain management therapy alone, and which variables may be associated with a better response to therapy. | Response will be measured after 24 weeks follow-up after the IPMT
  The therapies that will be analyzed are:
  * Fluoroscopically guided lumbar medial branch nerve radiofrequency denervation.
  * Fluoroscopically guided lumbar facet joint injection.
  * Fluoroscopically guided lumbar epidural corticosteroid injection.
  * Fluoroscopically guided caudal epidural corticosteroid injection.
  * Fluoroscopically guided pulsed radiofrequency of the lumbar dorsal root ganglion.
  * Fluoroscopically guided transforaminal epidural corticosteroid injection or lumbar selective root block.
Studying the association between main clinical diagnosis and the response to therapy, globally and stratified by single IPMT, after 4 weeks of the IPMT | Response will be measured after 4 weeks follow-up after the IPMT
  Main clinical diagnosis, response to therapy and IPMT performed are described separately as outcomes.
Studying the association between main clinical diagnosis and the response to therapy, globally and stratified by single IPMT, after 24 weeks of the IPMT | Response will be measured after 24 weeks follow-up after the IPMT
  Main clinical diagnosis, response to therapy and IPMT performed are described separately as outcomes.
Studying the satisfaction of the patients to the IPMT performed, after 24 weeks of IPMT | Satisfaction will be measured after 24 weeks follow-up after the IPMT
  Patient satisfaction will be assessed as two separate YES/NO questions:
  * Are you satisfied with the pain-relief obtained after you underwent the Interventional Pain Management Technique? (YES/NO answer).
  * Based on your experience, would you undergo the same treatment again? (YES/NO answer).
Studying the satisfaction of the patients to the IPMT performed, after 4 weeks of IPMT | Satisfaction will be measured after 4 weeks follow-up after the IPMT
  Patient satisfaction will be assessed as two separate YES/NO questions:
  - Are you satisfied with the pain-relief obtained after you underwent the Interventional Pain Management Technique? (YES/NO answer).
  Patient satisfaction will be assessed as two separate YES/NO questions:
  * Are you satisfied with the pain-relief obtained after you underwent the Interventional Pain Management Technique? (YES/NO answer).
  * Based on your experience, would you undergo the same treatment again? (YES/NO answer).
Studying the correlation of both scales (Numeric Rating Scale and Oswestry Disability Index) and patient satisfaction after 4 weeks of the IPMT | Response and satisfaction will be measured after 4 weeks follow-up after the IPMT
  Patient satisfaction will be assessed as two separate YES/NO questions:
  * Are you satisfied with the pain-relief obtained after you underwent the Interventional Pain Management Technique? (YES/NO answer).
  * Based on your experience, would you undergo the same treatment again? (YES/NO answer).
Studying the correlation of both scales (Numeric Rating Scale and Oswestry Disability Index) and patient satisfaction after 24 weeks of the IPMT | Response and satisfaction will be measured after 24 weeks follow-up after the IPMT
  Patient satisfaction will be assessed as two separate YES/NO questions:
  * Are you satisfied with the pain-relief obtained after you underwent the Interventional Pain Management Technique? (YES/NO answer).
  * Based on your experience, would you undergo the same treatment again? (YES/NO answer).
Studying the epidemiology and evolution of the pharmacological therapy of our population (Part I) | Drug therapy will be recorded at baseline
  Variable #1. Qualitative; is the patient taking any of the following medications (YES/NO for each treatment) at visit 0?:
  * Acetanomiphen.
  * Metamizole.
  * NSAID #1 (specify which).
  * NSAID #1 (specify which).
  * Gabapentine.
  * Pregabaline.
  * Tramadol.
  * Tapentadol.
  * Oxicodone.
  * Metadone.
  * Transdermic Fentanyl.
  * Transdermic Buprenorphine.
  * Amitriptiline.
  * Desipramine.
  * Nortriptiline.
  * Duloxetine.
  * Desvenlafaxine.
  * Paroxetine.
  * Citalopram.
  * Transdermic lidocaine.
  * Transdermic capsaicine.
  * Benzodiacepine (specify which).
  * Dexametasone.
  * Prednisone.
  * Hidrocodone.
  * Hidromorphone.
  * Oximorphine.
  * Minalcipram.
  * Bupropion.
  * Valproate.
  * Carbamazepine.
  * Lamotrigine.
  * Other (1) (specify which).
  * Other (2) (specify which).
  * Other (3) (specify which).
  Variable #2. Quantitative. 24 hour dose of each pharmacologic treatment the patient is taking at visit 0.
Studying the epidemiology and evolution of the pharmacological therapy of our population (Part II) | Drug therapy will be recorded at baseline; change in therapy will be recorded vs 4 weeks and vs 24 weeks.
  Variable #3. Qualitative. Is the patient taking any pharmacological treatment belonging to any of the following cathegories?:
  * NSAIDs, acetanomiphen, metamizole.
  * Opioids.
  * Oral opioids.
  * Minor opioids (tramadol, tapendatol, codeine)
  * Strong opioids.
  * Transdermic opioids.
  * Gabapentinoids.
  * Antidepressants.
  * Benzodiazepines.
  * Anticonvulsivants.
  Variable #4. Qualitative. Has it been any change in pharmacological treatment in the follow-up (baseline vs 4 weeks and vs 24 weeks) ; related to each pharmacological treatment)?:
  * Unchanged.
  * Higher dose.
  * Lower dose.
  * Treatment stopped.
  Variable #5. Qualitative. Why was the pharmacological treatment changed (baseline vs 4 weeks and vs 24 weeks) ?:
  * Clinical improvement.
  * Secondary effects.
  * Change for another pharmacological treatment.
Studying the safety and potential adverse reactions to IPMT. | Potential adverse reactions will be measured at the end of follow-up (after 24 weeks of the IPMT)
  Several cathegories:
  * Postdural puncture headache.
  * Infectious complication.
  * Epidural hematoma.
  * Neurologic damage.
  * Other (specify).
Studying the epidemiology of radiological findings in our population, and its association with the IPMT performed and the response to therapy after 4 weeks. | Response will be measured after 4 weeks follow-up after the IPMT
  Several cathegories or radiological findings:
  * Discopathy.
  * Herniated disk.
  * Central stenosis.
  * Lateral stenosis.
  * Radicular compression.
  * Spondyloarthrosis.
  * Spondylolisthesis.
  * Epidural fibrosis.
  * Reumatic inflammatory disease.
  * Vertebral compression fracture.
  * Scoliosis.
  * Other (specify).
Studying the epidemiology of radiological findings in our population, and its association with the IPMT performed and the response to therapy after 24 weeks. | Response will be measured after 24 weeks follow-up after the IPMT
  Several cathegories or radiological findings:
  * Discopathy.
  * Herniated disk.
  * Central stenosis.
  * Lateral stenosis.
  * Radicular compression.
  * Spondyloarthrosis.
  * Spondylolisthesis.
  * Epidural fibrosis.
  * Reumatic inflammatory disease.
  * Vertebral compression fracture.
  * Scoliosis.
  * Other (specify).
Studying the epidemiology of radiological findings in our population, and its association with clinical findings and clinical diagnosis. | Response will be measured after 24 weeks follow-up after the IPMT
  Several cathegories:
  * Discopathy.
  * Herniated disk.
  * Central stenosis.
  * Lateral stenosis.
  * Radicular compression.
  * Spondyloarthrosis.
  * Spondylolisthesis.
  * Epidural fibrosis.
  * Reumatic inflammatory disease.
  * Vertebral compression fracture.
  * Scoliosis.
  * Other (specify).
  Clinical findings are:
  * Fibromyalgia.
  * Failed back surgery syndrome.
  * Osteoporotic fracture.
  * Lumbar canal stenosis syndrome.
  * Irradiated pain to leg.
  * Arthrosis.
  * Inflammatory arthritis.
  * Oncologic condition.
  * Osteoporosis.
  Clinical diagnosis are defined as another outcome measure.
Analyzing the epidemiology of comorbidities (pain and not pain related) in our population: | Comorbidites will be recorded at baseline
  Comorbities that will be analyzed are:
  * Fibromyalgia.
  * Depression, anxiety and/or mixed axiety-depressive disorder.
  * Obesity.
  * Other chronic pain.
  * Failed back surgery syndrome.
  * Osteoporotic fracture.
  * Lumbar canal stenosis syndrome.
  * Irradiated pain to leg.
  * Diabetes Mellitus.
  * Arthrosis.
  * Inflammatory arthritis.
  * Oncologic condition.
  * Osteoporosis.
  * Substance abuse disorder.
Analyzing the demographical data of the study population. | Demographical data will be obtained at baseline
  Age, sex, marital status, working status at ethnic group and Medical Specialty that derivated the patient to our unit will be recorded at base line.
  * Working status: It will classified as: "active worker", "work sick leave", "studying", "retired person", "incapacitated to work" and "convict"
  * Marital status: It will classified as: "single", "unmarried partner", "married", "divorced" and "widowed".
  * Ethnic group: It will be classified as: "caucasic", "african"; "latin", "asiatic", "romany" and "other".
Studying the evolution in time of the response to the IPMT. | the response will be measured at +4weeks, +8weeks and +24 weeks
  Positive strong response, both strong (PSR) and moderate (PMR), as defined in "Primary outcomes" will be measured both at baseline vs 4 weeks follow-up, baseline vs 24 weeks follow-up and baseline vs 8 weeks follow-up.
  The evolution of the pain response will be studied; response and satisfaction will be measured at 4 different moments:
  * Baseline (prior to the performance of the IPMT).
  * 4 weeks after the IPMT is performed.
  * 8 weeks after the IPMT is performed.
  * 24 weeks after the IPMT is performed.
Charlson comorbidity index | Calculated at baseline
  Charlson comorbidity index will be calculated at baseline.
Pain syndrome | Pain syndrome is diagnosed at baseline
  Variable 1: presence of any of the following diagnosis:
  * Facet joint syndrome.
  * Vertebral crush fracture.
  * Discogenic pain.
  * Lateral lumbar canal stenosis.
  * Sacroiliac pain syndrome.
  * Central lumbar canal stenosis.
  * Failed back surgery syndrome.
  * None of the previous diagnosis. Variable n 2. Main pain syndrome, which is the one that motivates the IPMT.
  * Facet joint syndrome.
  * Vertebral crush fracture.
  * Discogenic pain.
  * Lateral lumbar canal stenosis.
  * Sacroiliac pain syndrome.
  * Central lumbar canal stenosis.
  * Failed back surgery syndrome.
  * None of the previous diagnosis.
  * There is no main pain syndrome: the patient has multiple pain diagnosis, and no single one prevails among the others. The IPMT is under a mixed therapeutic and diagnostic approach.
  Variable n3: number of pain syndromes present in the patient, of all the above.
Main operator of the IPMT | Measured 4 weeks after IPMT is performed
  Two cathegories:
  * Attending Pain Physician.
  * Anestesiology Resident.
Previous treatments, and success | Measured at baseline
  Variables n1 and n 2 are qualitative. Measured at visit 0.
  Variable n 1: the patient has undergone any of these treatments:
  * Back surgery.
  * Previous IPMT.
  * No IPMT.
  Variable n 2: subjective satisfaction of the patient:
  * Satisfied.
  * Not satisfied.
Numeric Rating Scale of pain at baseline | baseline
  The 11-point numerical pain rating scale (NRS) is a measure of pain in which patients rate their pain ranging from 0 (no pain) to 10 (worst imaginable pain). Validated in Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine 2005;30:1331-4.
Numeric Rating Scale of pain at 4 weeks after the IPMT is performed | 4 weeks after the IPMT is performed
  The 11-point numerical pain rating scale (NRS) is a measure of pain in which patients rate their pain ranging from 0 (no pain) to 10 (worst imaginable pain). Validated in Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine 2005;30:1331-4.
Numeric Rating Scale of pain at 8 weeks after the IPMT is performed | 8 weeks after the IPMT is performed
  The 11-point numerical pain rating scale (NRS) is a measure of pain in which patients rate their pain ranging from 0 (no pain) to 10 (worst imaginable pain). Validated in Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine 2005;30:1331-4.
Numeric Rating Scale of pain at 24 weeks after the IPMT is performed | 24 weeks after the IPMT is performed
  The 11-point numerical pain rating scale (NRS) is a measure of pain in which patients rate their pain ranging from 0 (no pain) to 10 (worst imaginable pain). Validated in Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine 2005;30:1331-4.
Oswestry Disability Index at baseline | baseline
  Original version 1 (1980), translated and adapted to Spanish (1995), validated.
Oswestry Disability Index at 4 weeks after the IPMT is performed | 4 weeks after the IPMT is performed
  Original version 1 (1980), translated and adapted to Spanish (1995), validated.
Oswestry Disability Index at 8 weeks after the IPMT is performed | 8 weeks after the IPMT is performed
  Original version 1 (1980), translated and adapted to Spanish (1995), validated.
Oswestry Disability Index at 24 weeks after the IPMT is performed | 24 weeks after the IPMT is performed
  Original version 1 (1980), translated and adapted to Spanish (1995), validated.
Clinical Frailty Scale at baseline | Obtained at baseline
  As described by Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I et al. A global clinical measure of fitness and frailty in elderly people. CMAJ 2005;173:489-95.
Previous treatments, and success | Mesured at baseline
  Variables n1 and n 2 are qualitative. Measured at visit 0.
  Variable n 1: the patient has undergone any of these treatments:
  * Back surgery.
  * Previous IPMT.
  * No IPMT.
  Variable n 2: subjective satisfaction of the patient:
  * Satisfied.
  * Not satisfied.
Interventional Pain Management Technique indicated at visit 0. | Baseline
  Several cathegories:
  * Fluoroscopically guided lumbar medial branch nerve radiofrequency denervation.
  * Fluoroscopically guided lumbar facet joint injection.
  * Fluoroscopically guided lumbar epidural corticosteroid injection.
  * Fluoroscopically guided caudal epidural corticosteroid injection.
  * Fluoroscopically guided pulsed radiofrequency of the lumbar dorsal root ganglion.
  * Fluoroscopically guided transforaminal epidural corticosteroid injection or lumbar selective root block.
Interventional Pain Management Technique performed. | Measured 4 weeks after the IPMT
  Several cathegories:
  * Fluoroscopically guided lumbar medial branch nerve radiofrequency denervation.
  * Fluoroscopically guided lumbar facet joint injection.
  * Fluoroscopically guided lumbar epidural corticosteroid injection.
  * Fluoroscopically guided caudal epidural corticosteroid injection.
  * Fluoroscopically guided pulsed radiofrequency of the lumbar dorsal root ganglion.
  * Fluoroscopically guided transforaminal epidural corticosteroid injection or lumbar selective root block.
Imaging modality | Baseline
  Qualitative:
  * MRI.
  * ST scan.
  * Lumbar x-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Garcia-Hernandez, Principal Investigator — Hospital General Universitario Gregorio Maranon; Ana Esther Lopez Perez, Study Chair — Hospital General Universitario Gregorio Maranon; Fernando Higuero-Cantonero, Principal Investigator — Hospital General Universitario Gregorio Maranon
Locations (1):
- Hospital General Universitario Gregorio Maranon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sivaganesan A, Chotai S, Parker SL, Asher AL, McGirt MJ, Devin CJ. Predictors of the efficacy of epidural steroid injections for structural lumbar degenerative pathology. Spine J. 2016 Aug;16(8):928-34. doi: 10.1016/j.spinee.2015.11.058. Epub 2015 Dec 9. PMID 26689476
- [Background] Manchikanti L, Buenaventura RM, Manchikanti KN, Ruan X, Gupta S, Smith HS, Christo PJ, Ward SP. Effectiveness of therapeutic lumbar transforaminal epidural steroid injections in managing lumbar spinal pain. Pain Physician. 2012 May-Jun;15(3):E199-245. PMID 22622912
- [Background] Cyteval C, Fescquet N, Thomas E, Decoux E, Blotman F, Taourel P. Predictive factors of efficacy of periradicular corticosteroid injections for lumbar radiculopathy. AJNR Am J Neuroradiol. 2006 May;27(5):978-82. PMID 16687527
- [Background] Park DY, Kang S, Park JH. Factors Predicting Favorable Short-Term Response to Transforaminal Epidural Steroid Injections for Lumbosacral Radiculopathy. Medicina (Kaunas). 2019 May 18;55(5):162. doi: 10.3390/medicina55050162. PMID 31109045